CLINICAL TRIAL: NCT02893787
Title: Study of Myocardial Function by Speckle Tracking After Cancer Treatment With Anthracyclines in Childhood
Acronym: SPECKLEANTHRA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9396
Record Dates: First submitted 2016-08-05; First posted 2016-09-09 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Myocardial Function; Echographic Parameters Obtaind by Speckle Tracking; Chilhood Cancers
Keywords: Speckle Tracking; Anthracyclines; Chilhood cancers; Myocardial function; Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients treated with anthracyclines in childhood
  Interventions: Other: Speckle Tracking Echocardiography
- Healthy volunteers
  Interventions: Other: Speckle Tracking Echocardiography

INTERVENTIONS:
Other: Speckle Tracking Echocardiography — Echocardiography analyses

SUMMARY:
The main goal of this study is to compare the values of echocardiographic parameters obtained by Speckle Traking analysis on myocardial function among patients under 18 years treated with anthracyclines in childhood, with healthy age and sex mached volunteers.

DETAILED DESCRIPTION:
Anthracyclines are major drugs in the treatment of childhood cancers. The main factor limiting their use is the occurrence of delayed cardiac toxicity, irreversible, in an dilated form of potentially fatal cardiomyopathy. This delayed cardiotoxicity secondary to the destruction of myocardial cells is histologically proven after administration of the first dose of anthracyclines. The main known risks factors for delayed cardiotoxicity are: the cumulative dose of anthracyclines, young age at the time of administration, and association with mediastinal radiotherapy. All pediatric protocols with anthracyclines therefore provide a prolonged cardiac monitoring.

However, there are no validated predictive early markers of progression to cardiomyopathy:

i) the standard echocardiography, routine surveillance method does not detect subclinical myocardial injury,

ii) the predictive value of biomarkers (ultrasensitive troponin, NT-pro-BNP) is controversial because of conflicting results.

Among the echocardiographic innovative techniques, myocardial strain imaging by speckle tracking echocardiography analyses via a software myocardial displacement of natural acoustic markers, and enables rapid evaluation, precise and objective of the segmental and global myocardial function, expressed as a percentage (strain) and speed of myocardial deformation (strain rate) by reference segment and by reference dimension (longitudinal, radial, circumferential).

Only four recent studies analysing the myocardic function in ST of the patients treated with anthracyclines in childhood (Yiu-fai, Cheung, Yu W, Poterucha) find unmatched and/or incomplete results, on a limited number of patients, but suggest the existence of alterations of the left ventricle the strain before the appearance of deteriorations of the fraction of ejection of the left ventricle (LVEF). None of these studies studied the strain of the right ventricle and none compared the data of the strain with the cardiac biomarkers.

Primary objective

Compare the values of echocardiographic parameters obtained by the technique of ST on myocardial function among patients under 18 years treated with anthracyclines in childhood, with healthy age and sex mached volunteers.

Secondary objectives

To compare conventional echocardiographic parameters and ST them in terms of deviation from the norm To assess the impact of known risk factors for cardiotoxicity with anthracyclines (cumulative dose, young age at administration, female association with mediastinal radiotherapy) on ultrasound parameters obtained by the technique of ST.

To evaluate the association between biomarkers for cardiotoxicity (ultrasensitive troponin and NT-pro-BNP) and echocardiographic parameters obtained by the technique of ST.

To correlate indices of Speckle Tracking methods to classical sonographic data

ELIGIBILITY:
Inclusion criteria:

* Patient treated between 0 and 18 with anthracyclines for malignancy
* Discontinuation of treatment with chemotherapy for over 1 year
* Patient in remission of his malignancy
* Lack of heart or lung disease associated
* No opposition patient and legal guardian
* Patient younger than 18 at the time of the study.

Exclusion criteria:

* Progressive malignant pathology.
* Cardiac, lung or muscle chronic diseases, etiology other than secondary to treatment with anthracyclines
* Refusal to participate in the study
* Poor echogenicity

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients under 18 years treated with anthracyclines in childhood and healthy age and sex mached volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Echocardiographic parameters obtained by Speckle Tracking | Immediat

CONTACTS AND LOCATIONS:
Overall Officials: Laure SAUMET, DR, Principal Investigator — Hôpital Arnaud de Villeneuve
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Amedro P, Vincenti M, Abassi H, Lanot N, De La Villeon G, Guillaumont S, Gamon L, Mura T, Lopez-Perrin K, Haouy S, Sirvent A, Cazorla O, Vergely L, Lacampagne A, Avesani M, Sirvent N, Saumet L. Use of speckle tracking echocardiography to detect late anthracycline-induced cardiotoxicity in childhood cancer: A prospective controlled cross-sectional study. Int J Cardiol. 2022 May 1;354:75-83. doi: 10.1016/j.ijcard.2022.02.012. Epub 2022 Feb 12. PMID 35167907